CLINICAL TRIAL: NCT05052216
Title: Development of a Wearable Point of Care Monitoring Device for Pediatric Obstructive Sleep Apnea
Status: Recruiting | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000224; 000224-CH
Record Dates: First submitted 2021-09-21; First posted 2021-09-22 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01-05

CONDITIONS: Pediatric Obstructive Sleep Apnea
Keywords: near-infrared spectroscopy (NIRS); tissue oxygenation; Polysomnography; Natural History

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NORM: healthy children
- OSA: children with obstructive sleep apnea

SUMMARY:
Background:

Obstructive sleep apnea (OSA) occurs when the blockage of the airway causes a person to stop breathing involuntarily for 10 seconds or more throughout the night during sleep. Pediatric OSA can be especially concerning and can have long-term effects. Researchers want to see how a monitoring device called near-infrared spectroscopy (NIRS) compares with the traditional techniques used in children s sleep studies.

Objective:

To learn about oxygen levels in the brain and limbs in children with and without sleep apnea using a wearable, point-of-care biosensor.

Eligibility:

Children aged 3-12 who have OSA and plan to receive treatment (OSA group) or who do not have OSA (NORM group).

Design:

Participants will be screened with a review of their medical records. If they have taken part in other NIH studies, that data will be reviewed as well.

Participants in the NORM group will have 1 overnight study visit. Those in the OSA group will have 2 overnight study visits.

Participants will do an overnight sleep study. They will have a physical exam and medical history. They will have a sleep study electroencephalography (EEG). For this, electrodes will be placed on their head. They will wear a gauze cap to keep the electrodes in place. Two NIRS probes made of a soft silicon will be placed on their forehead and arm. They will follow their normal bedtime routine. Their parent will stay overnight.

The OSA group will have a second study visit 2 weeks to 12 months after they start treatment for their sleep apnea. They will repeat the sleep study.

DETAILED DESCRIPTION:
Study Description:

This observational study will assess the sensitivity of near-infrared spectroscopy (NIRS) to hemodynamic events caused by pediatric obstructive sleep apnea (POSA). NIRS can provide a direct examination of brain oxygen saturation that traditional sleep study measurements are not able to capture and may be capable of better explaining health outcomes related to this disease. The purpose of this study is to characterize a wearable, point-of-care NIRS device that measures multiple physiological signals with a focus on cerebral and peripheral oxygenation in children with obstructive sleep apnea and to establish the relationship between traditionally measured parameters during sleep studies (polysomnography) and NIRS technologies. This study will be conducted in collaboration with the Sleep and Neurodevelopment Service at the NIH Clinical Center. Care will not be altered for any patients and this study will be purely observational with no significant risk added to any patient. We hypothesize that changes in NIRS signals of cerebral and peripheral tissue oxygenation due to apnea events will correlate with respiratory flow and oxygen saturation changes measured with PSG.

Objectives:

Primary Objective: Characterize cerebral oxygen saturation and peripheral tissue oxygen saturation during both normal sleep and sleep apnea events in children with respect to traditional polysomnography parameters.

Exploratory Objective 1: Characterize cerebral and peripheral tissue oxygen saturation before and after POSA treatment with respect to traditional polysomnography parameters.

Exploratory Objective 2: Characterize the dynamics of hemoglobin concentrations and tissue oxygenation during different sleep stages.

Exploratory Objective 3: Compare dynamics of cerebral and peripheral tissue oxygen saturation during apneic events in sleep state to a breath hold while subject is awake.

Endpoints:

Primary Endpoint: cerebral oxygen saturation (ScO2), peripheral tissue oxygen saturation (StO2), pulsatile oxygen saturation (SpO2), respiratory flow

Exploratory Endpoint 1: baseline and post-treatment ScO2, StO2, SpO2, AHI, respiratory flow

Exploratory Endpoint 2: baseline and post-treatment delta hemoglobin, delta deoxyhemoglobin, cerebral oxygen saturation

Exploratory Endpoint 3: ScO2, StO2 (during apnea and breath hold)

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Male or female, aged >=3 and <13 years
2. For NORM group: Children without OSA (AHI<2)
3. For OSA group: Children with OSA (AHI>=2)

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Children <3 years or >=13 years
2. Any chronic or acute medical condition that in the opinion of the investigators will interfere with overnight sleep study acquisition.
3. Any head injuries or physical conditions that in the opinion of the investigators would affect probe signal and contact.
4. For NORM group: Children with AHI>=2
5. For OSA group: Children with AHI<2

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: subjects enrolled in other sleep studies, subjects set to receive OSA treatment in the local area
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-08-25 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
ScO2, StO2 | Baseline
  peripheral tissue oxygen saturation (StO2), traditional polysomnography measures (SpO2, respiratory effort)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce J Tromberg, Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Not a clinical trial. This study serves as a pilot to evaluate and characterize a portable NIRS device for sleep research.

REFERENCES:
- [Background] Ullman N, Anas NG, Izaguirre E, Haugen W, Ortiz H, Arguello O, Nickerson B, Mink RB. Usefulness of cerebral NIRS in detecting the effects of pediatric sleep apnea. Pediatr Pulmonol. 2014 Oct;49(10):1036-42. doi: 10.1002/ppul.22962. Epub 2013 Dec 11. PMID 24339172
- [Background] Summerfelt ST, Selosse EJ, Reilly PJ, Trahanovsky WS. 1H-nuclear magnetic resonance spectroscopy of reducing-residue anomeric protons of pertrifluoroacetylated carbohydrates. Carbohydr Res. 1990 Aug 15;203(2):163-72. doi: 10.1016/0008-6215(90)80014-t. PMID 2276122
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000224-CH.html